CLINICAL TRIAL: NCT03243747
Title: Implementation of a Computer-based Questionnaire for Preoperative Evaluation in Anesthesia Ambulance
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Clinical Director of the Department of Anesthesiology and Operative Intensive Care Medicine Berlin (CCM, CVK), Charite University, Berlin, Germany
Other Study IDs: WAA
Record Dates: First submitted 2017-08-04; First posted 2017-08-09 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Patient Satisfaction; In-hospital Process Optimization
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preanesthetic evaluation is a clinical assessment process with purpose of increased patient safety. One focus is review of patient medical history to reduce perioperative morbidity and mortality as well as optimize the daily process in at anesthesia ambulance. The aim of that study is the development and implementation of a practical computer-based individualized and risk-adapted questionnaire for the daily routine

DETAILED DESCRIPTION:
The study was a step-by-step process. In the first investigation in 2013 the investigators included 50 patients and 81 patients in 2016. Questionnaires were identical in both testing stages for comparability. Practicability of a computer-based questionnaire on patient medical history, diagnosis as well as behavior guidelines was tested at anesthesia ambulance. Moreover, the investigators evaluated the user satisfaction with the help of a separate anonym paper-based questionnaire in 2013 as well as in 2016.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Patients who undergo a procedure in anaesthesia and elective surgery
* German speaking people

Exclusion Criteria:

* Emergency surgery
* American Society of Anesthesiologists (ASA) classification V and VI
* Patients with guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who undergo a procedure in anaesthesia and elective surgery at the Charité - Univeristätsmedizin Berlin, Campus Charité Mitte
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2016-10-14 (Actual)

PRIMARY OUTCOMES:
Utilization of computer-based questionnaire measured by duration time | Time in the outpatient clinic of anesthesia, an average of 1 hour
Number of assistance during filling-out in depending of age | Time in the outpatient clinic of anesthesia, an average of 1 hour

SECONDARY OUTCOMES:
Question 1: All in all I am content | Time in the outpatient clinic of anesthesia, an average of 1 hour
  User satisfaction evaluation by the help of a paper-based questionnaire
Question 2: The usability of tablet-pc is easy | Time in the outpatient clinic of anesthesia, an average of 1 hour
  User satisfaction evaluation by the help of a paper-based questionnaire
Question 3: My medical history is well determined | Time in the outpatient clinic of anesthesia, an average of 1 hour
  User satisfaction evaluation by the help of a paper-based questionnaire
Question 4: The phrasing of questions is clearly understandable | Time in the outpatient clinic of anesthesia, an average of 1 hour
  User satisfaction evaluation by the help of a paper-based questionnaire
Question 5: The total count of questions is acceptable | Time in the outpatient clinic of anesthesia, an average of 1 hour
  User satisfaction evaluation by the help of a paper-based questionnaire
Question 6: The complete duration time is acceptable | Time in the outpatient clinic of anesthesia, an average of 1 hour
  User satisfaction evaluation by the help of a paper-based questionnaire
Question 7: In the future, I would prefer digital questionnaires | Time in the outpatient clinic of anesthesia, an average of 1 hour
  User satisfaction evaluation by the help of a paper-based questionnaire
Question 8: In the future, I would prefer the questionnaire at home using internet. | Time in the outpatient clinic of anesthesia, an average of 1 hour
  User satisfaction evaluation by the help of a paper-based questionnaire. The evaluation was based on rating scale: 1=very good, 2=good, 3=satisfactory, 4=sufficient, 5=poor, 6=fail.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charité - Univsersitätsmedizin Berlin
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicne Berlin (CCM/CVK), Berlin, Germany

IPD SHARING:
Plan to Share IPD: No